CLINICAL TRIAL: NCT05680779
Title: Ultrasound-guided Percutaneous Neuromodulation in Patiens With Chronic Ankle Instability
Brief Title: Neuromodulation in Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, PhD Daniel Pecos-Martin, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEID/2022/2/031
Record Dates: First submitted 2022-12-23; First posted 2023-01-11 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNM group (Experimental): Subjects were treated once time. The technique consisted in the application of a square wave biphasic electrical current, with 10 Hz frequency, with 250 μs pulse width and the maximal torelable intensity to cause an exacerbated muscle contraction during ten seconds with a rest period of another ten seconds y total number of ten times. The subjects were lying in lateral decubitus. The common peroneal nerve was located with ultrasound (cross section) near to the peroneal head. After, an acupuncture needle (0,30mm x 30mm) was inserted in a long axis approach until the perineurium of the common peroneal nerve (in close proximity)
  Interventions: Other: ultrasound-guided percutaneous neuromodulation
- Control group (Other): Subjects were treated once time. The subjects were lying in lateral decubitus. The common peroneal nerve was located with ultrasound (cross section) near to the peroneal head. After, an acupuncture needle (0,30mm x 30mm) was inserted in a long axis approach until the perineurium of the common peroneal nerve (in close proximity). The needle remains in this location during 200 seconds without any electrical current.
  Interventions: Other: dry needling

INTERVENTIONS:
Other: ultrasound-guided percutaneous neuromodulation — It´s an intervention of physiotherapy
  Arms: PNM group
Other: dry needling — It´s an intervention of physiotherapy
  Arms: Control group

SUMMARY:
Ankle sprain is a common injury. Around 712,000 sprains occur every day in the world. It is estimated that they account for 45% of sports injuries, being the second part of the body that is most frequently injured in sports. Of the patients who suffer this injury, around 70% will develop chronic ankle instability, a situation that can cause residual pain, recurrent sprains, a feeling of lack of stability and decreased physical activity.

Two entities can be included in chronic ankle instability: mechanical instability, which involves movement of the joint beyond its physiological limit, and functional instability, which includes proprioceptive dysfunction, impaired neuromuscular control, postural control, and strength deficits.

Currently, the conservative treatment of these patients consists of neuromuscular training through the use of dynamic balance platforms, taping, joint mobilization, dry needling, and the use of plantar supports, balance training being the one that has shown the best result.

Ultrasound-guided percutaneous neuromodulation (PNM) is a recently used technique in the field of invasive physiotherapy that consists of applying a square wave biphasic electrical current through an acupuncture needle-like electrode that is place in close proximity to the nerve with ultrasound guidance. The aim of this study is to evaluate the effectiveness of PNM in ankle instability.

ELIGIBILITY:
Inclusion Criteria:

* Ankle instability

Exclusion Criteria:

* Subjects taking NSAIDs, analgesics or muscle relaxants
* Epilepsy
* Belonephobia or allergy to metals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-23 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Cumberland ankle instability tool | Change from Baseline up to three months
  The Cumberland ankle instability tool (CAIT) is a questionnaire that consists of 9 items, the maximum score of the questionnaire is 30 points, the lower the score obtained, the more severe the functional instability of the ankle. The Spanish version of the CAIT has high internal consistency (Cronbach's α00.766) and reliability (intraclass correlation coefficient 0.979, 95 % confidence interval (CI) 0.958-0.990).

SECONDARY OUTCOMES:
Byodex Balance System (BBS) | Change from Baseline up to 5 minutes
  The BBS is a platform designed to measure and record an individual´s ability to maintain stability under dynamic stress. It calculates a medial-lateral stability index (MLSI), anterior-posterior stability index (APSI), and an overall stability index (OSI) with reliability estimates of R= 0.92 (OSI), R = 0.89 (APSI), R= 0.93 (MLSI).
Electromyography muscle (EMG) | Change from Baseline up to 5 minutes
  Mdurance EMG system is valid tool to measure muscle activity during isokinetic contractions. It has shown an almost perfect Intraclass Correlation Coefficient>0.81.
stiffness tissue | Change from Baseline up to 5 minutes
  Myoton Pro is a device designed to measure and record Oscillation frequency (pitch), dynamic stiffness (stiffness), logarithmic decrement (elasticity), mechanical stress relaxation time and creep. It has shown an excellent reliability, Intraclass Correlation Coefficient 0.91-0.96 in all measures with the exception of elasticity 0.78-0.86

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, PhD, Study Chair — Alcala University
Locations (1):
- Physioterapy and Pain center research, Alcalá de Henares, Madrid, Spain